CLINICAL TRIAL: NCT01106950
Title: Adoptive Transfer of Haploidentical Natural Killer Cells to Treat Refractory or Relapsed AML MT2010-02
Brief Title: Haploidentical Natural Killer Cells to Treat Refractory or Relapsed Acute Myelogenous Leukemia (AML)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study drug (Ontak) no longer available
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010LS010; MT2010-02 (Other: Blood and Marrow Transplantation Program); 1003M79954 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Results first posted 2013-06-26 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Leukemia, Myelogenous, Acute
Keywords: acute myelogenous leukemia; primary acute myelogenous leukemia; secondary acute myelogenous leukemia; relapsed acute myelogenous leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — IL32 protein, human; fludarabine; fludarabine phosphate; Cyclophosphamide; denileukin diftitox; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated Patients (Experimental): Patients are treated with donor natural killer cells, fludarabine, cyclophosphamide, Denileukin diftitox, Donor lymphapheresis and IL-2.
  Interventions: Biological: Natural Killer Cells; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Denileukin diftitox; Procedure: Donor lymphapheresis; Drug: IL-2

INTERVENTIONS:
Biological: Natural Killer Cells — Given by infusion on Day 0. The product is T cell-depleted (CD3-) and B cell-depleted (CD19). Target dose for infusion is < or = 8 x 10^7 nucleated cells/kilogram.
Drug: Fludarabine — Administered as a 1 hour intravenous infusion once a day for 5 doses beginning on day -6.
  Other Names: Fludara
Drug: Cyclophosphamide — Administered as a 2 hour intravenous infusion with high volume fluid flush and mesna per institutional guidelines on day -5 and -4 one hour after fludarabine infusion. (Day -4 administration may be omitted if patient has had a transplant in the previous 4 months.)
  Other Names: Cytoxan
Drug: Denileukin diftitox — 12 ug/kg/day will be administered on day -1 and day -2 intravenously.
  Other Names: Ontak
Procedure: Donor lymphapheresis — Day -1 before planned NK cell infusion, the donor will undergo lymphapheresis (Removal of lymphocytes from donated blood, with the remainder of the blood retransfused into the donor).
Drug: IL-2 — Administered after NK cell infusion, 10 million units every other day for a total of 6 doses. (Patients weighing less than 45 kilograms will receive a dose of 5 million units/m^2 every other day for 6 doses).
  Other Names: Interleukin-2

SUMMARY:
This is a phase II therapeutic study of related donor HLA-haploidentical NK-cell based therapy after a high dose of fludarabine/cyclophosphamide with denileukin diftitox preparative regimen for the treatment of poor prognosis acute myelogenous leukemia (AML).

DETAILED DESCRIPTION:
Patients achieving a complete remission and neutrophil recovery (ANC > 500) for at least 4 weeks will be considered for allogeneic transplant to prolong remission (independent of this study).

All patients, including those who go on to transplant, will be followed to determine disease free survival, treatment related mortality, and time to relapse.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 2 years of age
* Meets one of the following disease criteria:

  * Primary acute myelogenous leukemia (AML) induction failure: no complete remission (CR) after 2 or more induction attempts
  * Relapsed acute myelogenous leukemia (AML): not in CR after 1 or more cycles of standard re-induction therapy. For patients > 60 years of age the 1 cycle of standard chemotherapy is not required if either of the following criteria is met:

    * relapse within 6 months of last chemotherapy
    * blast count < 30% within 10 days of starting protocol therapy
  * Secondary AML from myelodysplastic syndrome (MDS)
  * AML relapsed > 2 months after transplant who do not have the option of donor lymphocyte infusions (e.g. recipients of autologous or umbilical cord blood [UCB] transplants) Patients with prior central nervous system (CNS) involvement are eligible provided that it has been treated and CSF is clear for at least 2 weeks or magnetic resonance imaging (MRI) stable prior to enrollment. CNS therapy (chemotherapy or radiation) should continue as medically indicated during the study treatment.
* Available related HLA-haploidentical donor (3-5 of 6 HLA-A, B and C)
* Karnofsky Performance Status > 50% or Lansky Play score > 50
* Adequate organ function defined as:

  * Creatinine: ≤ 2.0 mg/dL (for pediatric patients - ClCr > 50 ml/min or age adjusted Cr)
  * Hepatic: Liver function tests (LFT's) < 5 x upper limit of institutional normal (ULN)
  * Pulmonary Function: oxygen saturation ≥ 90% on room air and pulmonary function >50% corrected Diffusion lung capacity for carbon monoxide (DLCO) and Forced expiratory volume in one second (FEV1) Oxygen saturation [>92%] can be used in child where pulmonary function tests (PFT's) cannot be obtained. (Testing required only if symptomatic or prior known impairment.)
  * Cardiac Function: Ejection fraction (EF) ≥ 40%, no uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Able to be off prednisone or other immunosuppressive medications for at least 3 days prior to natural killer (NK) cell infusion (excluding denileukin diftitox pre-meds)
* Women of child bearing potential must have a negative pregnancy test within 14 days prior to study registration and agree to use adequate birth control during study treatment.
* Voluntary written consent

Exclusion Criteria:

* Bi-phenotypic acute leukemia
* Transplant < 60 days prior to study enrollment
* New or progressive pulmonary infiltrates on screening chest x-ray or chest computated tomography (CT) scan that has not been evaluated with bronchoscopy, if feasible. Infiltrates attributed to infection must be stable/improving (with associated clinical improvement) after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections). Surgical resection waives any waiting requirements.
* Uncontrolled bacterial or viral infections - chronic asymptomatic viral hepatitis is allowed
* Pleural effusion large enough to be detectable on chest x-ray
* Known hypersensitivity to any of the study agents used
* Received investigational drugs within the 14 days before enrollment
* Known active CNS involvement

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Miller, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Bachanova V, Cooley S, Defor TE, Verneris MR, Zhang B, McKenna DH, Curtsinger J, Panoskaltsis-Mortari A, Lewis D, Hippen K, McGlave P, Weisdorf DJ, Blazar BR, Miller JS. Clearance of acute myeloid leukemia by haploidentical natural killer cells is improved using IL-2 diphtheria toxin fusion protein. Blood. 2014 Jun 19;123(25):3855-63. doi: 10.1182/blood-2013-10-532531. Epub 2014 Apr 9. PMID 24719405

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study entry was open to patients 2 years and older regardless of gender, race, or ethnic background.
Pre-assignment Details: Seventeen patients were enrolled, however, 2 patients did not receive Ontak (study drug) and were not included in the analysis.
Groups:
- Evaluable (Treated) Patients: Patients with acute myeloid leukemia (AML) are treated with donor natural killer cells, fludarabine, cyclophosphamide, Denileukin diftitox, Donor lymphapheresis and IL-2.
Period: Overall Study
Arm/Group | Evaluable (Treated) Patients
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Evaluable (Treated) Patients: Patients are treated with donor natural killer cells, fludarabine, cyclophosphamide, Denileukin diftitox, Donor lymphapheresis and IL-2.
Arm/Group | Evaluable (Treated) Patients
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 8
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (23.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With Successful Expansion of Natural Killer Cells After Infusion
Description: The primary objective of this study was to estimate the incidence of in vivo expansion of natural killer (NK) cells 14 days after infusion of an allogeneic donor product enriched for NK progenitors. Successful in vivo donor NK cell expansion was defined by measuring an absolute circulating donor-derived NK cell count of >100 cells/ul in the patient's peripheral blood 14 days after infusion.
Time Frame: Day 14
Measure: Number; unit: Percentage of patients
Groups:
- Evaluable (Treated) Patients: Patients with acute myeloid leukemia (AML) were treated with donor natural killer cells, fludarabine, cyclophosphamide, Denileukin diftitox, Donor lymphapheresis and IL-2.
Arm/Group | Evaluable (Treated) Patients
Number analyzed (Participants) | 15
Percentage of patients | 27

2. Secondary Outcome: Percent of Patients With Complete Remission of Disease
Description: Disease response was defined as complete remission (disease response) by morphologic criteria including <5% blasts in a moderately cellular or cellular marrow. Complete remission was also correlated with NK cell expansion in vivo, IL-15 levels and donor/recipient KIR B genotyping, and Treg depletion.
Time Frame: At least 4 weeks after last dose (28 days)
Measure: Number; unit: Percentage of patients
Arm/Group | Evaluable (Treated) Patients
Number analyzed (Participants) | 15
Percentage of patients | 53

3. Secondary Outcome: Percent of Patients With Disease Free Survival
Description: Number of patients alive and disease free at 6 months. The length of time after treatment ends that a patient survives without any signs or symptoms of that cancer or any other type of cancer. In a clinical trial, measuring the disease-free survival is one way to see how well a new treatment works.
Time Frame: Month 6
Measure: Number; unit: Percentage of patients
Arm/Group | Evaluable (Treated) Patients
Number analyzed (Participants) | 15
Percentage of patients | 33

4. Secondary Outcome: Percent of Patients With Incidence of Relapse
Description: Number of patients who have had a relapse(the return of disease after its apparent recovery/cessation) after obtaining a complete remission of their disease.
Time Frame: Month 6
Measure: Number; unit: Percentage of patients
Arm/Group | Evaluable (Treated) Patients
Number analyzed (Participants) | 15
Percentage of patients | 53

5. Secondary Outcome: Number of Patients With Treatment-Related Death
Description: Number of patients who died within the first 100 days of treatment due to toxicity.
Time Frame: Day 100
Measure: Number; unit: Percentage of patients
Arm/Group | Evaluable (Treated) Patients
Number analyzed (Participants) | 15
Percentage of patients | 13

6. Secondary Outcome: Percent of Patients With Natural Killer Cell Expansion Versus KIR Genotype Versus Treg Depletion
Description: Association between in vivo natural killer (NK) cell expansion and complete response without platelet recovery (CRp) with donor killer immunoglobulin-like (KIR) genotype and Treg depletion. In vivo donor NK cell expansion was correlated with regulatory T-cell (Treg) depletion as detected on flow cytometry.
Time Frame: Day 14
Measure: Number; unit: Percentage of patients
Groups:
- Evaluable (Treated) Patients (Expansion=No): KIR matched: Patients with acute myeloid leukemia (AML) were treated with donor natural killer cells, fludarabine, cyclophosphamide, Denileukin diftitox, Donor lymphapheresis and IL-2.
- Evaluable (Treated) Patients (Expansion=Yes): KIR mismatched: Patients with acute myeloid leukemia (AML) were treated with donor natural killer cells, fludarabine, cyclophosphamide, Denileukin diftitox, Donor lymphapheresis and IL-2.
Arm/Group | Evaluable (Treated) Patients (Expansion=No) | Evaluable (Treated) Patients (Expansion=Yes)
Number analyzed (Participants) | 7 | 8
Percentage of patients | 43 | 13

ADVERSE EVENTS:
Description: Due to chemotherapy as prep for the NK cell infusion, it is expected that all patients will experience severe depression of their blood counts and other related toxicities. Adverse event (AE) collection will focus on targeted AEs and unexpected AEs at specific time points in relation to the NK cell infusion and IL-2 injections.
Groups:
- Treated Patients: Patients with acute myeloid leukemia (AML) are treated with donor natural killer cells, fludarabine, cyclophosphamide, Denileukin diftitox, Donor lymphapheresis and IL-2.
Arm/Group | Treated Patients
Serious Adverse Events (participants affected / at risk) | 12/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Patients (N=15)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Blood disorder (Blood and lymphatic system disorders) | 5 (5)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1)
Hematologic toxicity - ANC<500 (Blood and lymphatic system disorders) | 1 (1)
Infusion related reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Typhilitis (Gastrointestinal disorders) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) — Grade 3
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 2
Lung Infection (Infections and infestations) | 1 (1) — Fungal pneumonia
Intracranial hemorrhage (Nervous system disorders) | 1 (1) — Possible fungal emboli
Encephalitis infection (Infections and infestations) | 1 (1) — CMV encephalitis and viremia
Infections and infestations- other (Infections and infestations) | 1 (1) — HHV6 positive bone marrow and blood cultures
Sepsis (Infections and infestations) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Patients (N=15)
Acute kidney injury - grade 1 (Renal and urinary disorders) | 2 (2)
Acute kidney injury - grade 2 (Renal and urinary disorders) | 2 (2)
Acute kidney injury - grade 3 (Renal and urinary disorders) | 2 (2)
Diffuse alveolar hemorrhage - grade 5 (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Gum/jaw pain - grade 2 (General disorders) | 4 (5)
Autoimmune disorder - grade 1 (Immune system disorders) | 15 (146)
Autoimmune disorder - grade 2 (Immune system disorders) | 2 (2)
Autoimmune disorder - grade 3 (Immune system disorders) | 9 (12)
Confusion - grade 4 (Nervous system disorders) | 1 (2)
Chills - grade 1 (Nervous system disorders) | 15 (130)
Chills - grade 2 (Nervous system disorders) | 14 (23)
Chills - grade 3 (Nervous system disorders) | 13 (28)
Dyspnea - grade 1 (Respiratory, thoracic and mediastinal disorders) | 15 (133)
Dyspnea - grade 2 (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Dyspnea - grade 3 (Respiratory, thoracic and mediastinal disorders) | 7 (15)
Dyspnea - grade 4 (Respiratory, thoracic and mediastinal disorders) | 5 (10)
Dyspnea - grade 5 (Respiratory, thoracic and mediastinal disorders) | 4 (15)
Edema - grade 1 (Blood and lymphatic system disorders) | 15 (113)
Edema - grade 2 (Blood and lymphatic system disorders) | 9 (36)
Edema - grade 3 (Blood and lymphatic system disorders) | 7 (28)
Edema - grade 4 (Blood and lymphatic system disorders) | 3 (8)
Headache - grade 1 (General disorders) | 2 (2)
Hypoxia - grade 1 (Respiratory, thoracic and mediastinal disorders) | 15 (147)
Hypoxia - grade 3 (Respiratory, thoracic and mediastinal disorders) | 5 (10)
Hypoxia - grade 4 (Respiratory, thoracic and mediastinal disorders) | 10 (20)
Hypoxia - grade 5 (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypertension - grade 1 (Cardiac disorders) | 14 (58)
Hypertension - grade 2 (Cardiac disorders) | 9 (42)
Hypertension - grade 3 (Cardiac disorders) | 13 (63)
Hypertension - grade 4 (Cardiac disorders) | 8 (20)
Hypotension - grade 1 (Cardiac disorders) | 15 (142)
Hypotension - grade 2 (Cardiac disorders) | 7 (20)
Hypotension - grade 3 (Cardiac disorders) | 6 (7)
Hypotension - grade 4 (Cardiac disorders) | 4 (12)
Infusion related reaction - grade 1 (Investigations) | 15 (156)
Infusion related reaction - grade 2 (Investigations) | 3 (4)
Infusion related reaction - grade 3 (Investigations) | 4 (4)
Fever - grade 1 (General disorders) | 15 (107)
Fever - grade 2 (General disorders) | 4 (4)
Fever - grade 3 (General disorders) | 3 (5)
Fever - grade 4 (General disorders) | 15 (62)
Pneumonitis/pulmonary infiltrates - grade 1 (Respiratory, thoracic and mediastinal disorders) | 15 (164)
Pneumonitis/pulmonary infiltrates - grade 3 (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Pneumonitis/pulmonary infiltrates - grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis/pulmonary infiltrates - grade 5 (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Rash/desquamation - grade 1 (Skin and subcutaneous tissue disorders) | 15 (152)
Rash/desquamation - grade 2 (Skin and subcutaneous tissue disorders) | 4 (9)
Rash/desquamation - grade 3 (Skin and subcutaneous tissue disorders) | 4 (7)
Rash/desquamation - grade 4 (Skin and subcutaneous tissue disorders) | 1 (13)
Abdominal distension - grade 2 (Gastrointestinal disorders) | 1 (1)
Bruising - grade 2 (Blood and lymphatic system disorders) | 1 (1)
Chest pain - grade 3 (General disorders) | 1 (1)
Blood disorder - grade 3 (Blood and lymphatic system disorders) | 1 (1)
Adult respiratory distress syndrome - grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Autoimmune disorder - grade 4 (Immune system disorders) | 1 (1)
Confusion - grade 3 (Nervous system disorders) | 1 (1)
Emesis - grade 3 (Gastrointestinal disorders) | 1 (1)
Heart failure - grade 4 (Cardiac disorders) | 1 (1)
Headache - grade 2 (General disorders) | 1 (1)
Headache - grade 4 (General disorders) | 1 (1)
Pneumonitis/pulmonary infiltrates - grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile neutropenia - grade 3 (Blood and lymphatic system disorders) | 1 (1)
Left ventricular systolic dysfunction - grade 3 (Cardiac disorders) | 1 (1)
Pneumonitis - grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intracranial hemorrhage - grade 2 (Vascular disorders) | 1 (1)
Lung infection - grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased creatinine - grade 2 (Endocrine disorders) | 1 (1)
Increased creatinine - grade 3 (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes